CLINICAL TRIAL: NCT02260050
Title: Bioequivalence of 20 mg of the New Formulation of WAL 801 CL Dry Syrup Compared to 20 mg of the Conventional Formulation of WAL 801 CL Dry Syrup Following Oral Administration in Healthy Male Volunteers (an Open-label, Randomised, Single-dose, 2x2 Crossover Study)
Brief Title: Bioequivalence of the New Formulation of WAL 801 CL Dry Syrup Compared to the Conventional Formulation of WAL 801 CL Dry Syrup in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 262.284
Record Dates: First submitted 2014-10-07; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- WAL 801 CL new formulation (Experimental)
  Interventions: Drug: WAL 801 CL dry syrup new formulation
- WAL 801 CL conventional formulation (Active Comparator)
  Interventions: Drug: WAL 801 CL dry syrup conventional formulation

INTERVENTIONS:
Drug: WAL 801 CL dry syrup new formulation
  Arms: WAL 801 CL new formulation
Drug: WAL 801 CL dry syrup conventional formulation
  Arms: WAL 801 CL conventional formulation

SUMMARY:
To establish the bioequivalence of the new formulation of WAL 801 CL dry syrup vs. the conventional formulation of WAL 801 CL dry syrup

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria:

  * Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR), body temperature (BT)), 12-lead ECG, clinical laboratory tests (including gastric acidity (GA) test)
  * No finding of clinical relevance
  * No evidence of a clinically relevant concomitant disease
* Age ≥ 20 and Age ≤ 35 years
* BMI ≥ 18.5 and BMI ≤ 25 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to Screening Phase and prior to Treatment Phase (Day -1 in Treatment period 1) in accordance with Japanese Good Clinical Practice (GCP)

Exclusion Criteria:

* Current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* History of surgery of gastrointestinal tract with the exception of appendectomy
* History of (and/or current) diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Current chronic or relevant acute infections
* History of hypersensitivity (including drug allergy) or current allergic disorders which are deemed relevant to the trial by the investigator or the sub-investigators; e.g. bronchial asthma, allergic rhinitis, atopic dermatitis and food allergy (excluding asymptomatic seasonal rhinitis/hay fever)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to drug administration and during Treatment Phase
* Use of any drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation, within 10 days prior to administration and during Treatment Phase
* Participation in Phase I trial of new chemical entities within 4 months prior to drug administration and during the trial, or in another clinical trial within 3 months prior to drug administration and during Treatment Phase
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking during hospitalization
* Alcohol abuse (more than 60 g/day) (confirmed by interview)
* Drug abuse (confirmed by interview)
* Whole blood donation (400 mL within 3 months or more than 100 mL within 4 weeks prior to drug administration or during the trial) or component blood donation (within 2 weeks prior to drug administration or during Treatment Phase)
* Excessive physical activities (within 48 hours prior to each treatment period and during hospitalisation)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2004-06; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to last measurable concentration (AUC0- tz) | up to 34 hours after drug administration
Maximum measured concentration of the analytes in plasma (Cmax) | up to 34 hours after drug administration

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 34 hours after drug administration
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | up to 34 hours after drug administration
Terminal rate constant of the analyte in plasma (λz) | up to 34 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | up to 34 hours after drug administration
Mean residence time of the analyte in the body after po administration (MRTpo) | up to 34 hours after drug administration
Number of patients with clinically significant findings in laboratory tests | up to 34 hours after last drug administration
Number of patients with clinically significant findings in physical examination | up to 34 hours after last drug administration
Number of patients with clinically significant findings in vital signs | Up to 34 hours after last drug administration
  blood pressure, pulse rate, body temperature
Number of patients with adverse events | Up to 48 hours after last drug administration